CLINICAL TRIAL: NCT06847867
Title: A Phase 2, Randomized, Open-label, Study of Momelotinib in Participants With Anemia Due to Low-risk Myelodysplastic Syndrome
Brief Title: A Study of Momelotinib in Participants With Low-risk Myelodysplastic Syndrome
Acronym: MIDAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 223584; 2024-519928-24 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Momelotinib; Low-risk Myelodysplastic Syndrome; MIDAS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1- Dose Optimisation: Momelotinib (Experimental)
  Interventions: Drug: Momelotinib
- Part 2- Dose Exploration: Momelotinib (Experimental)
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — Momelotinib will be administered.
  Other Names: GSK3070785

SUMMARY:
The goal of this clinical trial is to determine if momelotinib is safe and effective for people with low-risk myelodysplastic syndromes (LR-MDS). The trial will also examine how the body processes the drug. The study is comprised of two parts: Part 1: Participants will receive different doses of momelotinib to find the best dose by evaluating effectiveness in improving red blood cell transfusion requirements and safety. Part 2: Participants will receive dose selected from Part 1 to assess its impact on improving red blood cell transfusion requirements and safety in LR-MDS.

ELIGIBILITY:
Inclusion Criteria:

• Age ≥18 years or of legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent form (ICF).

* Documented diagnosis of MDS according to the World Health Organization classifications with an Revised International Prognostic Scoring System (IPSS-R) classification of very low, low, or intermediate risk disease, with an overall risk score ≤3.5.
* Received prior treatment with Erythropoiesis-stimulating agent (ESA) OR luspatercept for LR-MDS-related anemia that is relapsed/refractory to therapy. Participants intolerant to prior ESA or luspatercept will fulfill this inclusion criterion provided the definition below is met.

  - Refractory to prior treatment: documentation of loss of erythroid (E) response or never achieved HI-E response as defined by the IWG 2018 criteria.

  - Intolerant to prior treatment: documentation of reasons for discontinuation of prior ESA containing regimen, either as single agent or combination (e.g., G-CSF) or luspatercept due to intolerance or adverse event.
* Red blood cell transfusion dependence, defined as requiring an average of ≥4 units of Packed red blood cells (pRBC) transfused over an 8-week period during the 16 weeks preceding randomization. Documentation of a participant's transfusion policy during this 16-week period is required.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  a. Is a woman of non-childbearing potential (WONCBP). OR b. Is a woman of childbearing potential (WOCBP) and using a contraceptive method.
* Is capable of giving signed informed consent.
* Eastern Cooperative Oncology Group performance status ≤2.
* Adequate organ function.

Exclusion Criteria:

Prior treatment with the following with noted time periods:

1. Janus kinase (JAK)1/2 inhibitors; ACTRIIb IMiDs (iif ≤1 week of treatment received; provided last dose was ≥8 weeks from randomization
2. ACTRIIb receptor ligand trap other than luspatercept
3. Hypomethylating agents or other disease modifying agents (i.e., IMiDs) and immunosuppressive therapy for MDS
4. ESA within 4 weeks, or 8 weeks for long-acting ESA.
5. Growth factors (i.e., G-CSF, GM-CSF) within 4 weeks.
6. Luspatercept within 8 weeks.
7. Investigational agents within 4 weeks or 5 half-lives, whichever is longer.
8. Corticosteroids for treatment of the underlying disease within 28 days. Supportive care use of steroids for non-MDS indications may be used provided participant is on a stable dose equivalent to ≤10 mg prednisone per day.
9. Other active anti-MDS therapy not otherwise listed within 28 days or 5 half-lives whichever is longer.
10. Potent cytochrome P450 3A4 (CYP3A4) inducers, except for rifampin and rifampicin, within 14 days prior to the first dose of momelotinib.
11. Has received a live vaccine within 30 days. • Prior allogeneic or autologous stem cell transplant. • Has had any major surgery within 28 days prior to randomization. • Ongoing adverse reaction(s) from prior therapy that have not recovered to ≤Grade 1 or to the baseline status preceding prior therapy, except if the investigator, with the agreement of the sponsor, considers to be not clinically relevant for the tolerability of study intervention in the current clinical study.

    * MDS associated with del 5q cytogenetic abnormality.
    * Secondary MDS (i.e., MDS that is known to have arisen as the result of chemical injury, treatment with chemotherapy, and/or radiation for other diseases).
    * Known history of diagnosis of acute myeloid leukemia.
    * Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, gastrointestinal bleeding, or thalassemia.
    * Diagnosis of invasive malignancy or history of invasive malignancy other than the disease under study within the last 5 years, except as noted below:

<!-- -->

1. History of an invasive malignancy for which the participant was definitively treated, and in which the participant has been disease free for at least 2 years, and which, in the opinion of the principal investigator and medical monitor, is not expected to affect the evaluation of the effects of the study intervention on the currently targeted disease under study.
2. Curatively treated basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, and/or in situ breast cancer may be enrolled.
3. Incidental histologic finding of prostate cancer (T1a or T1b using the Tumor, nodes, metastasis [TNM] clinical staging system).

   * Uncontrolled intercurrent illness including, but not limited to:

a. Active uncontrolled infection (participants receiving outpatient antibacterial and/or antiviral treatments for infection that is under control or as infection prophylaxis may be included in the trial); or b. Significant active or chronic bleeding event ≥Grade 2 per Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) within 4 weeks prior randomization.

c. Uncontrolled acute and chronic liver disease (e.g., Child-Pugh score ≥10) OR has current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Any of the following conditions within 6 months prior to randomization:

1. Unstable angina pectoris.
2. Symptomatic congestive heart failure.
3. Uncontrolled cardiac arrhythmia. • QTc interval >480 milliseconds (msec) (corrected using Fridericia formula).

   • Psychiatric illness, social situation, or any other condition that would limit compliance with trial requirements or may interfere with the interpretation of study results, as judged by investigator or sponsor.

   • Presence of peripheral neuropathy ≥Grade 2 per CTCAE v5.0.

   • Known positive status for human immunodeficiency virus (HIV).

   • Hepatitis A, B, or C status as defined below:

a. Chronic active or acute viral hepatitis A. b. Active Hepatitis B infection indicated by the presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to the first dose of study intervention.

• Positive hepatitis C antibody test result at screening or within 3 months before the first dose of study intervention. Has any clinically significant gastrointestinal conditions or abnormalities that may alter absorption, e.g., uncontrolled nausea, vomiting, malabsorption syndrome or major resection of the stomach and/or bowels.

* Is unable to swallow and/or retain oral medications.
* Known contraindication or hypersensitivity to momelotinib and its metabolites, or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2029-03-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of participants with Red Blood Cells - transfusion independence (RBC-TI) for at least 12 weeks, rolling over 24 weeks | Up to 24 weeks
  RBC-TI defined as not requiring RBC transfusions (except in the case of clinically overt bleeding). Percentage of participants with RBC-TI will be measured for any consecutive 12-week interval over 24-week duration.
Part 1: Number of participants with Grade 3 Adverse events (AEs), AE leading to treatment discontinuation and AEs leading to dose modifications | Up to approximately 104 weeks
Part 1: Maximum plasma concentration (Cmax) of momelotinib and major metabolite of momelotinib (M21) | Up to 24 weeks
Part 1: Area under the plasma concentration versus time curve (AUC) of momelotinib and M21 | Up to 24 weeks
Part 2: Percentage of participants with ≥12 weeks of RBC-TI by the end of Week 24 | At week 24
  RBC-TI defined as not requiring RBC transfusions (except in the case of clinically overt bleeding). Percentage of participants with RBC-TI will be measured for any consecutive ≥12-week interval by the end of Week 24.

SECONDARY OUTCOMES:
Part 1: Percentage of participants with ≥12 weeks of RBC-TI by the end of Week 24 | At week 24
  RBC-TI defined as not requiring RBC transfusions (except in the case of clinically overt bleeding). Percentage of participants with RBC-TI will be measured for any consecutive ≥12-week interval by the end of Week 24.
Part 1: Number of participants with AEs, Serious adverse events (SAEs), AEs leading to treatment discontinuation, and AEs leading to dose modifications | Up to approximately 183 weeks
Part 1: Number of participants with AEs, SAEs, AEs leading to treatment discontinuation, and AEs leading to dose modifications by Severity | Up to approximately 183 weeks
Part 1: Number of participants with clinically significant changes in laboratory parameters | Up to approximately 183 weeks
Part 1: Number of participants with clinically significant changes in vital signs | Up to approximately 183 weeks
Part 1: Plasma concentration of momelotinib and M21 | Up to 24 weeks
Part 2: Percentage of participants with RBC-TI for ≥16 weeks by the end of Week 24 | At week 24
  RBC-TI defined as not requiring RBC transfusions (except in the case of clinically overt bleeding). Percentage of participants with RBC-TI will be measured for any consecutive ≥16-week interval by the end of Week 24.
Part 2: Percentage of participants with ≥1.5 grams per deciliter (g/dL) increase in hemoglobin | Up to 48 weeks
Part 2: Percentage of participants with RBC-TI for ≥24weeks by the end of Week 48 | At week 48
  RBC-TI defined as not requiring RBC transfusions (except in the case of clinically overt bleeding). Percentage of participants with RBC-TI will be measured for any consecutive ≥24-week interval by the end of Week 48
Part 2: Number of participants with hematologic improvement (HI-E) response per International Working Group (IWG) 2018 criteria | Up to 24 weeks
  HI-E response is measured based on the combined incidence of: Low transfusion burden (LTB) patients defined as absence of any transfusion for ≥ 8 consecutive weeks. High transfusion burden (HTB) patients: minor response defined as reduction by ≥ 50% of red blood cell (RBC) units for ≥ 8 consecutive weeks. Major response defined as absence of RBC transfusions for ≥ 8 consecutive weeks or longer up to 24 weeks
Part 2: Time to RBC-TI by Weeks 24 and 48 | Up to Weeks 24 and 48
  Time to RBC-TI defined as the time from the first dose of study intervention until the first date of TI (absence of RBC transfusion requirement).
Part 2: Number of participants with AEs, SAEs, AEs leading to treatment discontinuation, AEs leading to dose modifications | Up to approximately 183 weeks
Part 2: Number of participants with AEs, SAEs, AEs leading to treatment discontinuation, AEs leading to dose modifications by severity | Up to approximately 183 weeks
Part 2: Number of participants with clinically significant changes in laboratory parameters | Up to approximately 183 weeks
Part 2: Number of participants with clinically significant changes in vital signs | Up to approximately 183 weeks
Part 2: Plasma concentration of momelotinib and M21 | Up to 24 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.